CLINICAL TRIAL: NCT04525469
Title: Feasibility Trial of Narrative Exposure Therapy (NET) for Posttraumatic Stress Disorder (PTSD) During Pregnancy
Acronym: NET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Natalie Stevens, Research Director, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18111901-IRB01
Record Dates: First submitted 2020-08-13; First posted 2020-08-25 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Post Traumatic Stress Disorder; Perinatal; Pregnancy; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative Exposure Therapy (Experimental): NET is a fully-manualized evidence-based treatment for PTSD. Participants will receive 6 weekly 60-minute individual sessions of NET.
  Interventions: Behavioral: Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — NET involves: 1) diagnostic interview and psychoeducation, 2) laying out the Lifeline, 3) NET therapy sessions (constructing the trauma narrative in context of the life course), 4) final session rituals. Laying out the Lifeline (using rope or string) allows participants to take a bird's eye view of the events of their life using simple items such as flowers to represent positive events and stones to represent traumatic events. The focus of NET sessions is to encourage participants to describe the details of traumas and integrating the "cold" memories (i.e., facts) with the "hot" memories (e.g., cognitions, emotions, physiological feelings, and sensory information). The therapist makes notes after each session narrating the details of the traumas ("stones") and reads this at the beginning of each subsequent session. Final session rituals involve re-reading the trauma narrative, hopes for the future, and laying out the final Lifeline placing flowers for hopes and wishes for the future.
  Other Names: NET

SUMMARY:
Posttraumatic stress disorder (PTSD) affects up to 35% of pregnant trauma survivors. Moreover, prenatal PTSD rates are up to 4 times higher among communities of color compared to white populations. PTSD during pregnancy has been linked to an increased risk of adverse perinatal and infant health outcomes and may even contribute to racial disparities in adverse perinatal outcomes. Although front-line treatments exist for PTSD, treatment research that specifically focus on pregnancy are extremely limited. Clinical studies examining the safety, acceptability, feasibility, and efficacy of treatments for PTSD during pregnancy are virtually non-existent. Thus, pregnant individuals with PTSD, particularly within low-income communities of color, are a vulnerable and underserved group in need of effective treatment approaches for their distress. Investigators propose to conduct a feasibility and acceptability study of a PTSD treatment, Narrative Exposure Therapy (NET), in a sample of pregnant individuals with PTSD in which low-income people of color are highly represented.

Aim 1: The purpose of Aim 1 will be to examine feasibility. Investigators will evaluate the recruitment and assessment procedures.

Aim 2: The purpose of Aim 2 will be to examine acceptability. Investigators will evaluate participant feedback of the NET intervention.

Aim 3: The purpose of Aim 3 will be to examine the proportion of participants demonstrating clinically meaningful reduction in PTSD and perinatal depression symptoms from pre- to post-treatment.

Investigators will aim to enroll up to 30 participants; participation will last up to ten months. Data sources will include questionnaires, electronic medical records, and qualitative feedback interviews.

With this study, investigators aim to fill a critical gap in knowledge of how to safely and effectively treat PTSD among a vulnerable and underserved population (i.e., perinatal individuals of color).

DETAILED DESCRIPTION:
Investigators will conduct a feasibility and acceptability study of Narrative Exposure Therapy (NET) to treat up to 30 pregnant trauma survivors with clinically-significant symptoms of PTSD.

Up to 100 participants will be recruited with the aim of enrolling 30 participants in NET. Pregnant patients will be recruited from Rush OB/GYN resident training clinics. The racial/ethnic composition of patients served at these clinics (>70% ethno-racial minorities) will ensure that participants of color will be highly represented. Methods of recruitment include NET brochures that will be placed in the clinic's waiting rooms, OB/GYN physicians and nurse referring patients with a known history of trauma, and a 2-item screening measure -- the PTSD Checklist, Civilian Version (PCL-2) -- at the patient's initial OB appointment to facilitate recruitment.

Following initial referral, the study team will conduct a brief phone screen to ensure basic eligibility criteria are met, describe the study purpose, and schedule eligible participants for an initial study session (week 0). During the initial visit participants will sign informed consent and complete self-report measures (week 1 of the study) - after which they will then be enrolled in the intervention (weeks 1-6 of the study). Participants will complete post-treatment self-report measures and treatment evaluation measures at 1 week and 1-month following their last NET session (week 7 and week 10, respectively), and again at 1-month postpartum. The participant will also be invited to complete a qualitative feedback interview upon completion of the intervention (or early withdrawal from intervention).

Participants will be compensated for completion of all assessments and study components.

Due to the Coronavirus/COVID-19 pandemic, all study activities will be conducted via telephone or telehealth.

Schedule of Activities:

* Week 1: Consent and Pre-Intervention Clinical AND NET Session 1 Consent Session/Pre-Intervention Clinical interview

  1. Informed Consent: If patients are interested in participating in this study, they will undergo the informed consent procedure. A trained clinician with experience working with trauma survivors will verbally review the informed consent document.
  2. Interview and Self-Report Measures:
  3. Participation in Treatment while enrolled in the study: Patients may be in or seek psychological or psychiatric treatment and still enroll in the study, as long as they are not undergoing exposure therapy. If patients indicate that they are already or wish to seek such treatment, they will be asked to provide consent for study personnel to contact their mental health provider to obtain this single piece of information, as well as whether or not they are being prescribed anti-psychotics (which is a reason for study exclusion)
* NET Session 1

  1. For each weekly session, the content of each session will be taken from the NET manual, a developed manualized treatment. The NET manual can be accessed here: https://www.psychologytools.com/category/narrative-exposure-therapy-net/
* Weeks 2-6: Sessions 2-6 of NET

  1. Participants will also complete self-report measures before the beginning of each NET session via REDCap.
* 1 Week Post-treatment: Post-treatment Evaluation
* 1 Month Post-treatment 10: Post-treatment Evaluation
* 1 Month Postpartum: Follow-up Evaluation
* Qualitative Feedback Interview (upon completion of the intervention or early withdrawal from intervention)

ELIGIBILITY:
Inclusion:

* 18 years of age or older
* Fluent in English
* History of a DSM-V PTSD criterion A trauma at least 3 months prior to current pregnancy (a person has experienced, witnessed, or been confronted with an event or events that involve actual or threatened death or serious injury, or threat of physical integrity to oneself or others)
* A score of 33 or higher on the PTSD Checklist for the DSM-V with Life Events Checklist for DSM-5 and Criterion A.

Exclusion:

* Current manic or psychotic symptoms or primary psychotic diagnosis
* Serious cognitive impairment
* Concurrent psychotherapy
* Unstable dose of psychotropic medications (must be stable for 6 weeks)
* Serious medical complications of pregnancy (e.g., pre-eclampsia, HELLP syndrome, diagnosed fetal anomaly or death, threatened preterm birth, hospitalization for hypertensive disorders of pregnancy, unstable diabetes, premature rupture of membranes, preterm labor)
* Significant suicidal ideation
* Current legal actions related to trauma
* Patient will be 27 gestational weeks or more at the time of the eligibility session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility via recruitment rate | Screening to enrollment (Week 1)
  Investigators will compute the number of phone screens conducted, number of eligibility sessions completed, and number of subjects enrolled to obtain participant enrollment rates.
Feasibility via retention rate (sessions completed/dropout rate) | Week 1 (NET Session 1) to Week 6 (NET Session 6)
  Investigators will calculate the mean number of sessions attended and the dropout rate, recording reason for drop out, such as participants' desire to withdraw from the NET treatment vs. medical complications of pregnancy or early delivery.
Feasibility via retention rate (completion of follow-up questionnaires) | 1 Week Post-treatment (Post-treatment Evaluation), 1 Month Post-treatment (Post-treatment Evaluation), 1 Month Post-partum (Follow-up Evaluation)
  Investigators will calculate the mean number of follow-up questionnaires completed.
Acceptability of the NET intervention via participant satisfaction | 1 Week Post-treatment (Post-treatment evaluation)
  Investigators will compute mean ratings of satisfaction (adapted Client Satisfaction Questionnaire).
Acceptability of the NET intervention via participant expectancy | Week 1 (NET Session 1) , Week 2, Week 3, Week 4, Week 5, Week 6 (NET Sessions 6)
  Investigators will compute mean ratings of expectancy via feasibility and acceptability questionnaires.
Acceptability of the NET intervention via perceived benefit | 1 Week Post-treatment (Post-treatment evaluation), 1 Month Post-treatment (post-treatment evaluation), 1 Month Postpartum (follow-up evaluation)
  Investigators will compute mean ratings of perceived benefit via post-treatment evaluations.
Acceptability of the NET intervention via qualitative feedback | Upon study completion (up to 10 months) or upon early withdrawal from intervention
  Primary outcome will include qualitative feedback regarding aspects of the NET intervention and its acceptability during pregnancy and in preparation for the transition to parenthood via a study-developed qualitative interview.
Change in Symptoms of PTSD | Week 1 (NET Session 1), 1 Week Post-treatment (Post-treatment evaluation), 1 Month Post-treatment (post-treatment evaluation), 1 Month Postpartum (follow-up evaluation)
  Investigators will use the Posttraumatic Check List for DSM-5 (PCL-5), a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD.

SECONDARY OUTCOMES:
Change in Symptoms of Perinatal Depression | Week 1 (NET Session 1), 1 Week Post-treatment (Post-treatment evaluation), 1 Month Post-treatment (post-treatment evaluation), 1 Month Postpartum (follow-up evaluation)
  Investigators will use the Edinburgh Postnatal Depression Scale (EPDS), a 10-item self-report measure for depression screening in the perinatal period.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevens NR, Miller ML, Soibatian C, Otwell C, Rufa AK, Meyer DJ, Shalowitz MU. Exposure therapy for PTSD during pregnancy: a feasibility, acceptability, and case series study of Narrative Exposure Therapy (NET). BMC Psychol. 2020 Dec 9;8(1):130. doi: 10.1186/s40359-020-00503-4. PMID 33298159